CLINICAL TRIAL: NCT04632355
Title: After the First and Second Wave in Italy: What Effects of Musculoskeletal Pain Did the Covid-19 in Patients Who Have Hospital Care?
Brief Title: Musculoskeletal Pain in Patients With Covid-19 Who Have Hospital Care
Acronym: Covid19-Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: Covid19-Pain
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: Covid19; Pain; musculoskeletal
MeSH Terms: conditions — COVID-19; Pain | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — This interview will be conducted to collecting all outcomes about musculoskeletal pain in COVID-19 survivors
  Other Names: COVID-19 survivors

SUMMARY:
Worldwide, the COVID-19 pandemic continues to grow. Although COVID-19 mainly affects the lungs and internal organs, musculoskeletal injury from this disease was reported with the presentation of marked elevation in creatine kinase and lactate dehydrogenase levels. Patients with post-acute COVID-19 are considered patients with a post-intensive syndrome (PICS) that results in loss of functional independence.

In the physical and rehabilitation medical field, various modalities with therapeutic exercise can be used to manage pain by a physical therapist and psychiatrist.

Pain management is particularly important during the COVID-19 pandemic because of the reduced accessibility to hospitals and medical resources.

DETAILED DESCRIPTION:
The COVID-19 survivors with pain symptoms will participated. In this phase, a face-to-face interview will be conducted to collecting all outcomes about pain.

ELIGIBILITY:
Inclusion Criteria:

* Recovered from COVID-19 infection.
* COVID-19 survivors after hospitalization.
* Musculoskeletal pain.

Exclusion Criteria:

* Participants will be excluded also if they score greater than 6 points on the Beck Depression Inventory (BDI) or more than 30 points in the State Trait Anxiety Inventory (STAI), dementia and not Italian speaking due to the high level of language skills required for questionnaires and quantitative sensory testing.
* Psychiatric or neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who had been recovered from COVID-19 infection, that is, COVID-19 survivors after hospitalization in the abovementioned Hospitals of Italy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported Version of the Leeds Assessment of Neuropathic Symptoms and Signs | Baseline
  the characterization of the pain. Total of 24. > 11 neuropathic pain.
PainDETEC | Baseline
  the characterization of the pain
EuroQol-5D | Baseline
  To measure quality of life, grade ranging from 0 (the worst possible health status) to 100 (the best possible health status)
The Hospital Anxiety and Depression Scale | Baseline
  To measure psychological status. 0-7 = Normal; 8-10 = Borderline abnormal (borderline case), 11-21 = Abnormal (case)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge H Villafañe, Principal Investigator — Fondazione Don Carlo Gnocchi
Locations (1):
- Jorge Hugo Villafañe, Milan, Italy

REFERENCES:
- [Background] Pedersini P, Corbellini C, Villafane JH. Italian Physical Therapists' Response to the Novel COVID-19 Emergency. Phys Ther. 2020 Jul 19;100(7):1049-1051. doi: 10.1093/ptj/pzaa060. No abstract available. PMID 32280973
- [Background] Pancera S, Galeri S, Porta R, Pietta I, Bianchi LNC, Carrozza MC, Villafane JH. Feasibility and Efficacy of the Pulmonary Rehabilitation Program in a Rehabilitation Center: CASE REPORT OF A YOUNG PATIENT DEVELOPING SEVERE COVID-19 ACUTE RESPIRATORY DISTRESS SYNDROME. J Cardiopulm Rehabil Prev. 2020 Jul;40(4):205-208. doi: 10.1097/HCR.0000000000000529. PMID 32609464